CLINICAL TRIAL: NCT00144313
Title: Persistence of Antibody and Response to Booster of a Recombinant Hepatitis B Vaccine in Children Who Responded to a Primary Course of 2.5µg Recombinant Hepatitis B Vaccine as Infants
Brief Title: VaxTeen Hepatitis B Vaccine Booster Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Alaska Native Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCID-4127; U50/CCU022279-01
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-09

CONDITIONS: Hepatitis
Keywords: vaccine; hepatitis B; immune memory
MeSH Terms: conditions — Hepatitis; Hepatitis B | interventions — Hepatitis B Vaccines

INTERVENTIONS:
Biological: hepatitis B vaccine

SUMMARY:
The purpose of this study is to determine immune status of adolescents who responded to a primary series of recombinant hepatitis B vaccine given at birth and to assess their response to a booster dose of vaccine.

DETAILED DESCRIPTION:
In the 1970s, Alaska Natives had the highest rate of hepatitis B virus (HBV) infection in the US. Because of this, routine vaccination for all Alaska Native infants beginning at birth was implemented in 1985. Hepatitis B vaccination programs have resulted in significant declines in acute and chronic HBV infections among Alaska Natives, with virtually no new chronic infections observed among the vaccinated cohort. Since 1991, the American Academy of Pediatrics (AAP) and the Advisory Committee on Immunization Practices (ACIP) have recommended hepatitis B vaccination for all infants, preferably beginning at birth. Beginning vaccination during infancy prevents childhood acquisition of HBV, and provides immunity against HBV before individuals reach an age where they may be at increased risk of exposure due to high-risk behaviors (i.e., sexual activity and drug use) or occupation.

The success of this vaccination strategy is contingent on the vaccine being able to induce long-lasting protection. The duration of protection conferred by hepatitis B vaccination initiated at birth is not firmly established. Over 95% of vaccinees in clinical studies develop a response to the three-dose primary hepatitis B vaccination series, defined as the development of antibody to hepatitis B virus surface antigen (anti-HBs) to concentrations greater than10 milliInternational Units per milliliter (mIU/mL) in blood. Within 5-10 years after the primary series, anti-HBs concentrations decline and for many vaccinees, concentrations will fall below 10mIU/mL, or even below detectable levels.

However, despite low anti-HBs concentrations, HBV infections (as measured by the presence of markers of infection such as hepatitis B surface antigen [HBsAg] or antibody to hepatitis B core antigen [anti-HBc]) are rare in persons who have been shown to respond to the primary vaccine series. Continued protection against HBV infection in these children is likely provided by immune memory cells generated at the time of the primary series. An immunologic memory response (also termed an anamnestic response) can be evaluated by measuring the effect of an additional (booster) dose of hepatitis B vaccine. An anamnestic response is generally defined as a rapid (within 14-30 days) two-fold or greater increase in the anti-HBs titer to at least 20mIU/mL. This signifies that immune memory cells capable of generating a rapid rise in anti-HBs are still functional and would protect against HBV infection. Blood tests that can identify memory B cells that are specific for vaccine antigens are now available, and could be used to provide additional evidence of immune memory.9

Although there is good evidence that the immunologic memory for HBsAg exceeds the persistence of measurable antibodies, few studies have examined lasting protection (>10 years) against HBV infection in a low-risk population vaccinated at birth with recombinant vaccine.10 Most studies demonstrating long term protection from infection and persistent immune memory despite low anti-HBs concentrations have been performed among children living in areas where HBV infection is endemic, or whose mothers had chronic HBV infection (i.e., children at high risk of perinatal or childhood HBV infection). Studies conducted among Alaska Native children have demonstrated that "low-risk" children (i.e., infants who were born to HBsAg-negative mothers with no HBsAg-positive persons living in their households) also have concentrations of anti-HBs that fall below 10mIU/mL during later childhood. In a cohort of 36 children known to have responded to a recombinant vaccine series starting at birth, none retained levels of anti-HBs ≥ 10mIU/mL at 7.5 years of age. In addition, three of these children failed to exhibit an anamnestic response to a booster dose given at an average age of 7.5 years.

At the present time, neither measurement of anti-HBs concentrations nor booster dose(s) are recommended for low-risk children after the hepatitis B vaccine primary series given during infancy. Low-risk Alaska Native children who received recombinant hepatitis B vaccination starting at birth are now reaching adolescence, a period when the risk of HBV infection through sexual transmission or transmission by injecting drug use is more likely to occur. More information is needed to determine if protection against HBV infection among children entering adolescence is adequate or if booster dose(s) might be necessary.

The specific objectives are as follows:

Primary

1. To determine anti-HBs concentrations among adolescents aged 11-14 years old who responded to a primary series of recombinant hepatitis B vaccine initiated at birth.
2. To assess the anti-HBs response to a booster dose of recombinant hepatitis B vaccine among adolescents who have been previously shown to respond to a primary series of recombinant hepatitis B vaccine initiated at birth.
3. To determine whether specific immune memory cells are present among the study cohort members.

Secondary

1. To correlate the response to a booster dose of hepatitis B vaccine with

   1. initial response to the primary series
   2. concentration of anti-HBs and age at time of a booster dose.
2. To document side effects in persons receiving a fourth dose of hepatitis B vaccine.
3. To determine the proportion of children who received and responded to a primary vaccine series in infancy who subsequently became infected with HBV as demonstrated by the presence of anti-HBc and/or HBsAg.

ELIGIBILITY:
Inclusion Criteria:

* Eligible children are those who received the 2.5 µg/dose three-dose series of Recombivax HB® with the first dose having been given during the first week of life and the series completed by 9 months. All children were born to HBsAg
* negative mothers, had no HBsAg-positive persons living in their households at the time of immunization, and had a minimum of one serologic specimen prior to the age of 18 months with results indicating an anti-HBs concentration of ≥10mIU/mL.

Exclusion Criteria:

* Receipt of a fourth dose of any hepatitis B vaccine
* History of allergic reaction after receiving hepatitis B vaccine or hypersensitivity to any components of the hepatitis B vaccine used for the booster dose
* History of hepatitis B virus infection
* Existence of disease known to affect the immune system (e.g., HIV, AIDS, SCID, chronic renal disease, cancer)
* Current or recent (within 6 months) receipt of immunomodulatory therapy (e.g., systemic corticosteroids, chemotherapy) or blood products

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2005-08; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
anti-HBs concentration

SECONDARY OUTCOMES:
side effects
anti-HBc and/or HBsAg following primary vaccine series in infancy

CONTACTS AND LOCATIONS:
Overall Officials: Laura L Hammitt, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- CDC Arctic Investigations Program, Anchorage, Alaska, United States